CLINICAL TRIAL: NCT01123720
Title: To Understand the Impacts of Internationalize Medical Services on Local People Seeking Medical Care, and to Establish Responsive Management Mechanism
Brief Title: The Impact of Internationalize Medical Services to localPeople Seeking Medical Care
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Taiwan College of Healthcare Executives (Unknown)
Responsible Party: Lan-Chin Lu, Taipei Medical University WanFang Hospital
Other Study IDs: 099M031
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Administrative Staff in Hospital of Taiwan

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recently The Department of Health of Taiwan has launched the "Internationalize Medical Services Flagship Program", expecting to promote Taiwan's high-quality of medical services to the international market, and anticipating "customers stroll in, medical services walked out".

In order to avoid expansion of this program might alienate the rights and best interests of local people seeking medical services, therefore, this research project is a join effort of experts to form an advisory counsel; by collecting most current international medical services data; then using both qualitative and quantitative questionnaires to investigate whether by implementation of internationalize medical services will cause great impact on local people.

To study the various of insurance income of health care organization after they promote international medical services; and to understand the impact of assess to medical care and quality of medical services to local people due to internationalize medical services.

The last through advisory counsel, to make specific recommendations on mechanism of management and to set evaluation of indicators to monitor international health care, to avoid edge out local people the right of seeking medical care to ever happened, and to aid future planning of policy and implementation.

DETAILED DESCRIPTION:
The main objectives of this study are:

1. To understand the impact from internationalize medical services to local People seeking medical care, and the impact to management of health care organization, make specific recommendations for assessment, management mechanisms and measurable indicators, and aid future planning of policy and implementation.
2. To avoid expanding the flagship program of internationalization of medical services might jeopardize local people's right to seek medical care, assess the impact to local people after the program implemented.

ELIGIBILITY:
Inclusion Criteria:

* Administrative staff in Hospital
* Hospital provide the internationalize medical services

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Administrative staff in Hospital of Taiwan
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lan-Chin Lu, Principal Investigator — Taipei Medical University WanFang Hospital